CLINICAL TRIAL: NCT01927107
Title: Effects of Probiotics Mixture to Standard Diet Therapy in Obese Children
Brief Title: Effects of Probiotics in Obese Children
Acronym: Prob-esity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Eskisehir Osmangazi University (Other)
Responsible Party: Principal Investigator, Ener Cagri DINLEYICI, Associate Professor in Pediatrics, Eskisehir Osmangazi University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Prob-esity
Record Dates: First submitted 2013-08-16; First posted 2013-08-22 (Estimated); Last update posted 2017-07-28 (Actual); Status verified 2017-07

CONDITIONS: Obesity
Keywords: probiotics; obesity; oxidative stress
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Probiotic mixture (Active Comparator): Probiotic mixture including Lactobacillus acidophilus (4.3x108CFU/per sachet), Lactobacillus rhamnosus (4.3x108CFU/ per sachet), Bifidobacterium bifidum (4.3x108CFU/ per sachet), Bifidobacterium longum (4.3x108CFU/ per sachet), Enterococcus faecium (8.2x108CFU/ per sachet, per oral daily for 30 days in addition to standard approach
  Interventions: Dietary Supplement: Probiotics mixture
- Control (Active Comparator): Standard diet therapy
  Interventions: Dietary Supplement: Probiotics mixture

INTERVENTIONS:
Dietary Supplement: Probiotics mixture — Comparison of probiotic mixture in addition to standard diet therapy vs. standart diet therapy

SUMMARY:
The global obesity epidemic presents an unprecedented challenge to the public health worldwide. The factors associated with obesity are complex, and include health behaviors, such as eating habits and daily physical activity, and broader social, environmental and biological determinants that influence these health behaviors. The intestinal microbiota has several beneficial functions related to host health and accumulating evidence indicates that the gut microbiota plays a significant role in the development of obesity, obesity-associated inflammation and insulin resistance. Experimental studies reveal a shift in the abundance of Bacteroidetes and Firmicutes. Presumably, obesity affects the diversity of the gut microbiota and, probably, the way individuals harvest energy from nutrients. Differences in community composition, functional genes and metabolic activities of the gut microbiota appear to distinguish lean vs obese individuals, suggesting that gut 'dysbiosis' contributes to the development of obesity and/or its complications.

Recent studies have suggested some beneficial effects of probiotics and/or prebiotics on obesity and metabolic syndrome in adults; such experience is limited in children and adolescents. The aim of this study was to evaluate potential effects of add-on probiotics to standard therapy on anthropometric measurements, lipid profile and oxidative stress parameters in children.

DETAILED DESCRIPTION:
he global obesity epidemic presents an unprecedented challenge to the public health worldwide. The factors associated with obesity are complex, and include health behaviors, such as eating habits and daily physical activity, and broader social, environmental and biological determinants that influence these health behaviors. The intestinal microbiota has several beneficial functions related to host health and accumulating evidence indicates that the gut microbiota plays a significant role in the development of obesity, obesity-associated inflammation and insulin resistance. Experimental studies reveal a shift in the abundance of Bacteroidetes and Firmicutes. Presumably, obesity affects the diversity of the gut microbiota and, probably, the way individuals harvest energy from nutrients. Differences in community composition, functional genes and metabolic activities of the gut microbiota appear to distinguish lean vs obese individuals, suggesting that gut 'dysbiosis' contributes to the development of obesity and/or its complications.

Recent studies have suggested some beneficial effects of probiotics and/or prebiotics on obesity and metabolic syndrome in adults; such experience is limited in children and adolescents. The aim of this study was to evaluate potential effects of add-on probiotics to standard therapy on anthropometric measurements, lipid profile and oxidative stress parameters in children.

ELIGIBILITY:
Inclusion Criteria:

* Children with obesity according to anthropometric measurements with appropriate weight for age

Exclusion Criteria:

* coexistence of secondary obesity, malignancy, immune deficiency, collagen vascular diseases, congenital anomalies, neurological findings, children with receiving concomitant any drugs related chronic condition or antibiotics. Children with exogenous obesity who have also insulin resistance and /or hypertension were also excluded

Ages: 5 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 120 (Actual)
Dates: Start 2012-04; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Obesity related anthropometric measurements | 30th days
  Change of obesity related anthropometric measurements including weight, body mass index, upper arm circumference, tirceps skinfold thickness, waist and hip circumference

SECONDARY OUTCOMES:
Evaluation of biochemical indices and oxidative stress | 30th days
  Serum total cholesterol level, serum triglyceride level, serum LDL-C levels, serum HDL-C levels, serum total anti-oxidant capacity levels, serum total oxidative stress level
Safety | 30th days
  Side effects related with probiotic use: nausea, vomiting, other GIS disturbances, rash

CONTACTS AND LOCATIONS:
Overall Officials: Ener C Dinleyici, MD, Principal Investigator — Eskisehir Osmangazi University